CLINICAL TRIAL: NCT01810029
Title: A Randomized Controlled Trial of Stress Reduction in the Secondary Prevention of Coronary Heart Disease in African Americans
Brief Title: A Trial of Stress Reduction in the Secondary Prevention of Coronary Heart Disease in Blacks
Acronym: CCR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maharishi International University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director, Center for Natural Medicine and Prevention, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1RC1HL100386-01 (NIH)
Record Dates: First submitted 2012-04-18; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: transcendental meditation; cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiac Rehabilitation; Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac Rehabilitation plus Transcendental Meditation (Experimental): a standard validated cardiac rehabilitation program plus a standard validated stress reduction component, the Transcendental Meditation program
  Interventions: Behavioral: Cardiac Rehabilitation plus Transcendental Meditation
- Cardiac Rehabilitation (Active Comparator): This control is a standard Cardiac Rehabilitation without a stress reduction technique
  Interventions: Behavioral: Cardiac Rehabilitation plus Transcendental Meditation

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation plus Transcendental Meditation — The stress reduction intervention, Transcendental Meditation program is added on to the standard cardiac rehabilitation programs for patients with documented coronary artery disease
  Other Names: TM technique, TM program, Transcendental Meditation

SUMMARY:
The overall hypothesis of this study is that a cardiac rehabilitation program with meditation will be more effective than cardiac rehabilitation alone in improving blood flow through the diseased coronary arteries in African Americans. For this purpose, 56 African American men and women with coronary heart disease will be randomly assigned either to standard cardiac rehabilitation plus the Transcendental Meditation program or to standard cardiac rehabilitation alone. The treatment period will be 12 weeks in length.

DETAILED DESCRIPTION:
The overall objective of this study is to conduct a randomized controlled trial to determine the efficacy of cardiac rehabilitation with and without a structured, standardized, and validated stress reduction component in the secondary prevention of coronary heart disease (CHD) in African Americans. In this phase II trial, 56 African American men and women with established CHD will be randomly allocated either to standard cardiac rehabilitation with formal stress reduction training using the Transcendental Meditation program or to standard cardiac rehabilitation alone. The intervention period will be 12 weeks. At baseline and posttest, subjects will be tested by quantitative Positron Emission Tomography (PET) for myocardial perfusion and ischemia. Secondary outcomes comprise physiological, behavioral and psychosocial risk factors for CHD. The field site will be Columbia University Medical Center and the coordinating center will be MUMRI-Center for Natural Medicine and Prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age: No limitations
3. CHD documented by medical history of at least one of the following: a.acute myocardial infarction (MI) within the preceding 12 months b.coronary artery bypass surgery (CABG) c. percutaneous coronary intervention (PCI, PTCA)d. chronic stable angina
4. Written informed consent

Exclusion Criteria:

1. noncardiac life threatening illness
2. Severe cognitive impairment or physical disability
3. History of major psychiatric disorder, i.e. psychosis, dementia, or substance abuse disorder within the past year.
4. Left ventricular ejection fraction less than 40%
5. Conditions that may be a contraindications to PET perfusion imaging with adenosine stress testing, including unstable angina or myocardial infarction in the past week, aortic stenosis, uncontrolled hypertension, uncontrolled atrial or ventricular arrhythmias, second-degree or higher atrio-ventricular block in the absence of a functioning pacemaker, baseline hypotension (systolic blood pressure < 90 mm Hg), severe obstructive lung disease or decompensated heart failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
coronary blood flow as measured by PET | 12 weeks

SECONDARY OUTCOMES:
blood pressure, behavioral risk factors (diet, exercise, substance use) and psychosocial stress factors (depression, social support, general well-being) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University
Locations (1):
- Columbia University Medical Center, Dept of Cardiology, New York, New York, United States

REFERENCES:
- [Derived] Bokhari S, Schneider RH, Salerno JW, Rainforth MV, Gaylord-King C, Nidich SI. Effects of cardiac rehabilitation with and without meditation on myocardial blood flow using quantitative positron emission tomography: A pilot study. J Nucl Cardiol. 2021 Aug;28(4):1596-1607. doi: 10.1007/s12350-019-01884-9. Epub 2019 Sep 16. PMID 31529385